CLINICAL TRIAL: NCT05136989
Title: Psychiatry and Individual Liberties: a Study of Institutions Characterized by a Reduced Use of Coercion
Acronym: (PLAID-Care)
Status: Recruiting | Type: Observational
Sponsor: Centre Hospitalier Universitaire de Saint Etienne (Other)
Collaborators: L'École Nationale des Solidarités, de l'Encadrement et de l'Intervention Sociale (ENSEIS) (Unknown)
Responsible Party: Sponsor
Other Study IDs: IRBN1372021/CHUSTE
Record Dates: First submitted 2021-11-16; First posted 2021-11-30 (Actual); Last update posted 2024-03-12 (Actual); Status verified 2024-03

CONDITIONS: Psychiatric Hospitalization
Keywords: Psychiatry; Reduction of coercion; Interviews; Observations; Sociology; Nursing

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Professionals from the seven least coercive facilities: Volunteer professionals selected on the basis of their experience in reducing the use of coercion.
  Interventions: Behavioral: Individual and collective semi-structured interviews; Behavioral: Observations out in the services
- Voluntary ex-patients: Voluntary ex-patients who were hospitalized in these establishments in the two years preceding the survey and whose condition is stabilized
  Interventions: Behavioral: Individual semi-structured interviews with ex-patients

INTERVENTIONS:
Behavioral: Individual and collective semi-structured interviews — Individual and collective semi-structured interviews will be performed with professionals to identify levers (practices, knowledge, tools, regulations) which, at the level of services and establishments, enable the development of a policy of less recourse to coercion
  Groups: Professionals from the seven least coercive facilities
Behavioral: Individual semi-structured interviews with ex-patients — Individual semi-structured interviews will be performed with ex-patients in order to gather their experiences in the seven institutions concerned and to better understand the impact of their hospitalization in these institutions on their lives
  Groups: Voluntary ex-patients
Behavioral: Observations out in the services — Observations will be carried out in the services in order to measure the gap between rhetoric and practice, and to observe the effective implementation of lesser use practices
  Groups: Professionals from the seven least coercive facilities

SUMMARY:
Psychiatric establishments show significant disparities in terms of coercion: while some use it frequently, others use it only exceptionally. This project aims at a better understanding of the less coercive establishments, which are currently little investigated and whose study may allow to identify the levers of a psychiatry more respectful of individual liberties.

DETAILED DESCRIPTION:
This study aims precisely at understanding the history of less coercive establishments, and at identifying the knowledge as well as the forms of organization, coordination and cooperation that are developed there. To do so, it will consist of an inventory of establishments and practices based on the analysis of scientific literature, and an intensive study of seven less coercive establishments (four establishments on the French national territory, three establishments in the Auvergne-Rhône-Alpes region). The study of these institutions and their environment, which mobilizes nursing research and sociology, is based on a methodological approach combining interviews with professionals and users, observations in the institutions and services, a documentary method, and analysis of data from the RIM-P, the SAE, and the institutions' databases.

ELIGIBILITY:
Inclusion Criteria:

* Professionals who worked in one of the seven establishments identified
* Ex-patients who were hospitalized in these establishments in the two years preceding the survey and whose condition is stabilized

Exclusion Criteria:

* People who refused to participate to the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The research focuses mainly on care and support professionals, administrative and management staff, and users of seven establishments or poles identified as less coercive (three establishments in the Auvergne-Rhône-Alpes region, and four establishments on the national territory).
Sampling Method: Non-Probability Sample
Enrollment: 98 (Estimated)
Dates: Start 2021-12-01 (Actual); Primary Completion 2024-06 (Estimated); Study Completion 2024-06 (Estimated)

PRIMARY OUTCOMES:
understand the history of less coercive institutions | Baseline from 24 months
  identify and characterize the presence of tools, knowledge, rules, organizational specificities and collaborations in the territories allowing for less recourse to coercion.

SECONDARY OUTCOMES:
Analysis of professionals' satisfaction | Baseline from 24 months
  Analysis interview responses
Analysis of ex-patients' satisfaction | Baseline from 24 months
  Analysis interview responses.
Analysis of the impact on care pathway | Baseline from 24 months
  Analysis interview responses.
Analysis of the impact on career paths | Baseline from 24 months
  Analysis interview responses.

CONTACTS AND LOCATIONS:
Overall Officials: Sébastien SAETTA, PhD, Principal Investigator — CHU de Saint-Etienne
Locations (1):
- CHU Saint Etienne, Saint-Etienne, France